CLINICAL TRIAL: NCT05789615
Title: Letermovir Prophylaxis for Cytomegalovirus Infection in Haploidentical Allogeneic Hematopoietic Cell Transplant Recipients: Single-center Real-world Data in China
Brief Title: Letermovir Prophylaxis for CMV Infection in Haplo-HSCT Recipients: Single-center Data in China
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SOOCHOW-WXJ-2022-366
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: CMV Infection; Hematopoietic Stem Cell Transplantation
Keywords: Letermovir; Cytomegalovirus Infection; Haploidentical HSCT
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 200 haplo-HSCT recipients who are CMV seropositive: The study consists 200 cases CMV-R+ adult (>18 years) recipients of haplo-HCT. All patients will receive letermovir prophylaxis. Consider a simple interim analysis of the experimental group could be arranged after 150 patients are enrolled if necessary.
  Supportive care is provided by institutional standards of care (e.g., acyclovir for herpes simplex virus and varicella zoster virus prevention).
  Letermovir prophylaxis is started on day 0 or no longer than 28 days after transplantation. During the study period, letermovir 480 mg PO/IV once daily (or 240 mg per day in patients taking cyclosporine) was administered from day 0 to day +100 post-HCT.
  CMV monitoring and preemptive therapy were performed according to local protocol. Plasma CMV viral load (VL) is monitored by quantitative CMV PCR, starting on day +7 and continued weekly until week 6, then every 2-4 weeks for months until week 24.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Letermovir has achieved excellent therapeutic benefits globally but is still in its infancy in China. Letermovir obtained an implied license for a clinical trial in June 2020, and in November 2020, Letermovir submitted and accepted four new drug marketing applications in China, including injection and tablet formulations. On December 31, 2021, the China National Medical Products Administration (NMPA) approved letermovir for cytomegalovirus (CMV) seropositive adult recipients undergoing allogeneic hematopoietic stem cell transplantation (HSCT) [R+] prevention of cytomegalovirus infection and cytomegalovirus disease. The commercial launch of letermovir is estimated to be in August 2022.

SUMMARY:
In the 30 years of fighting CMV infection, the mortality rate among HSCT patients has significantly reduced. Now, the focus is on improving the prognosis of HSCT patients and preventing CMV infection. The emergence of letermovir has provided a new opportunity in this regard. Letermovir, the only drug approved for CMV infection prevention in HSCT patients, works by inhibiting the CMV DNA terminase complex. Phase III studies have shown that letermovir significantly reduces CMV infection and all-cause mortality after HSCT, without increasing myelosuppression or nephrotoxicity. Real-world studies have further confirmed its efficacy in reducing CMV infection rates and antiviral use. Letermovir's global success has not yet been fully realized in China, where it is still in its early stages of use.

DETAILED DESCRIPTION:
Letermovir achieved excellent therapeutic outcomes globally but is still developing in China. It received an implied license for clinical trials in June 2020, followed by marketing applications in November 2020. In December 2021, it was approved by the China National Medical Products Administration (NMPA) for preventing CMV infection and disease in CMV seropositive adult recipients undergoing allogeneic hematopoietic stem cell transplantation (HSCT). Letermovir's commercial launch in China is expected in August 2022. Given that over 90% of the Chinese population is CMV seropositive, determining whether CMV prevention is necessary based solely on serology is insufficient. The growing use of haploidentical stem cell transplantation (haplo-SCT) in China, particularly using the Beijing protocol for GVHD prevention, increases CMV risk. However, limited data exists on the efficacy of CMV prophylaxis for haplo-SCT patients in China. A real-life study assessing the efficacy, resistance, and tolerability of letermovir in this patient group is essential to guide CMV management strategies, particularly for high-risk CMV R+ haploidentical transplant recipients. This prospective study aims to evaluate letermovir's real-life impact on efficacy, resistance, tolerability, and CMV-related morbidity and mortality in China.

ELIGIBILITY:
Inclusion Criteria:

* Haplo-SCT candidate (adult) who has decided to primary transplant and is willing to participate in the study.
* The haplo-SCT candidate (adult) should be CMV seropositive recipients.

Exclusion Criteria:

* CMV-seronegative patient receiving a negative CMV donor graft.
* Patients having active CMV DNAemia at the time of letermovir initiation.
* Patient having signed the informed consent but not grafted.
* Patient recruited in a clinical study on an anti-CMV trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consists 200 cases CMV-R+ adult (>18 years) recipients of haplo-HCT. All patients will receive letermovir prophylaxis.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant CMV infection | at Week 14 following haplo-SCT
  Defined as CMV DNAemia leading to preemptive treatment or presence of CMV disease using classificatory criteria published by the Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. CMV DNA threshold for initiation of preemptive therapy at our center is viral load >500 copies/mL or above on two consecutive tests.

SECONDARY OUTCOMES:
Incidence of clinically significant CMV infection | through Week 24 following haplo-SCT
  Defined as CMV DNAemia leading to preemptive treatment or presence of CMV disease using classificatory criteria published by the Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. CMV DNA threshold for initiation of preemptive therapy at our center is viral load >500 copies/mL or above on two consecutive tests.
Incidence of CMV DNAemia and CMV disease | through Week 14 and Week 24 following haplo-SCT
  CMV DNAemia refers to the presence of CMV DNA in the blood. CMV disease refers to the organ dysfunction caused by an active CMV infection, such as the lungs, liver, and retina.
Incidence of the resistant or refractory CMV infection | through Week 24 following haplo-SCT
  Resistant or refractory CMV infection occurs if CMV levels rise by 1 log after 2 weeks of treatment or remain positive after 4 weeks.
Incidence of serious adverse event leading to interruption of treatment | through Week 24 following haplo-SCT
  Serious adverse events refers to events that require stopping the treatment to ensure patient safety.
Incidence of CMV-related disease mortality | through Week 24 following haplo-SCT
  Death resulting directly or indirectly from complications of a CMV infection, often involving severe organ damage in the lungs, liver, or other organs.
Incidence of all-cause mortality and non-relapse mortality | through Week 24 following haplo-SCT
  All-cause mortality refers to deaths from any cause, while non-relapse mortality refers to deaths caused by factors other than the recurrence or relapse of the original disease or condition.
Incidence of CMV-associated morbidity | through Week 24 following haplo-SCT
  CMV-associated morbidity refers to organ damage, delay engraftment, acute or chronic GVHD occurrence, or other infectious diseases caused by CMV.
Incidence of rehospitalization | through Week 14, Week 24 following haplo-HSCT
  The frequency or rate at which patients are readmitted to the hospital within a specified period following their discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojin Wu, Prof., Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Styczynski J. Who Is the Patient at Risk of CMV Recurrence: A Review of the Current Scientific Evidence with a Focus on Hematopoietic Cell Transplantation. Infect Dis Ther. 2018 Mar;7(1):1-16. doi: 10.1007/s40121-017-0180-z. Epub 2017 Dec 4. PMID 29204910
- [Background] Green ML, Leisenring W, Xie H, Mast TC, Cui Y, Sandmaier BM, Sorror ML, Goyal S, Ozkok S, Yi J, Sahoo F, Kimball LE, Jerome KR, Marks MA, Boeckh M. Cytomegalovirus viral load and mortality after haemopoietic stem cell transplantation in the era of pre-emptive therapy: a retrospective cohort study. Lancet Haematol. 2016 Mar;3(3):e119-27. doi: 10.1016/S2352-3026(15)00289-6. Epub 2016 Feb 20. PMID 26947200
- [Background] Tomblyn M, Chiller T, Einsele H, Gress R, Sepkowitz K, Storek J, Wingard JR, Young JA, Boeckh MJ; Center for International Blood and Marrow Research; National Marrow Donor program; European Blood and MarrowTransplant Group; American Society of Blood and Marrow Transplantation; Canadian Blood and Marrow Transplant Group; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America; Association of Medical Microbiology and Infectious Disease Canada; Centers for Disease Control and Prevention. Guidelines for preventing infectious complications among hematopoietic cell transplantation recipients: a global perspective. Biol Blood Marrow Transplant. 2009 Oct;15(10):1143-238. doi: 10.1016/j.bbmt.2009.06.019. No abstract available. PMID 19747629
- [Background] Akahoshi Y, Kimura SI, Inamoto Y, Seo S, Muranushi H, Shimizu H, Ozawa Y, Tanaka M, Uchida N, Kanda Y, Katayama Y, Shiratori S, Ota S, Matsuoka KI, Onizuka M, Fukuda T, Atsuta Y, Murata M, Terakura S, Nakasone H. Effect of Cytomegalovirus Reactivation With or Without Acute Graft-Versus-Host Disease on the Risk of Nonrelapse Mortality. Clin Infect Dis. 2021 Aug 2;73(3):e620-e628. doi: 10.1093/cid/ciaa1871. PMID 33341890
- [Background] Hakki M, Aitken SL, Danziger-Isakov L, Michaels MG, Carpenter PA, Chemaly RF, Papanicolaou GA, Boeckh M, Marty FM. American Society for Transplantation and Cellular Therapy Series: #3-Prevention of Cytomegalovirus Infection and Disease After Hematopoietic Cell Transplantation. Transplant Cell Ther. 2021 Sep;27(9):707-719. doi: 10.1016/j.jtct.2021.05.001. PMID 34452721
- [Background] Razonable R. Direct and indirect effects of cytomegalovirus: can we prevent them? Enferm Infecc Microbiol Clin. 2010 Jan;28(1):1-5. doi: 10.1016/j.eimc.2009.07.008. Epub 2009 Dec 21. No abstract available. PMID 20022410
- [Background] Goodrich JM, Mori M, Gleaves CA, Du Mond C, Cays M, Ebeling DF, Buhles WC, DeArmond B, Meyers JD. Early treatment with ganciclovir to prevent cytomegalovirus disease after allogeneic bone marrow transplantation. N Engl J Med. 1991 Dec 5;325(23):1601-7. doi: 10.1056/NEJM199112053252303. PMID 1658652
- [Background] Boeckh M, Nichols WG. The impact of cytomegalovirus serostatus of donor and recipient before hematopoietic stem cell transplantation in the era of antiviral prophylaxis and preemptive therapy. Blood. 2004 Mar 15;103(6):2003-8. doi: 10.1182/blood-2003-10-3616. Epub 2003 Nov 26. PMID 14644993
- [Background] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658
- [Background] Su Y, Stern A, Karantoni E, Nawar T, Han G, Zavras P, Dumke H, Cho C, Tamari R, Shaffer B, Giralt S, Jakubowski A, Perales MA, Papanicolaou G. Impact of Letermovir Primary Cytomegalovirus Prophylaxis on 1-Year Mortality After Allogeneic Hematopoietic Cell Transplantation: A Retrospective Cohort Study. Clin Infect Dis. 2022 Sep 14;75(5):795-804. doi: 10.1093/cid/ciab1064. PMID 34979021
- [Background] Derigs P, Radujkovic A, Schubert ML, Schnitzler P, Schoning T, Muller-Tidow C, Hegenbart U, Schonland SO, Luft T, Dreger P, Schmitt M. Letermovir prophylaxis is effective in preventing cytomegalovirus reactivation after allogeneic hematopoietic cell transplantation: single-center real-world data. Ann Hematol. 2021 Aug;100(8):2087-2093. doi: 10.1007/s00277-020-04362-2. Epub 2020 Dec 3. PMID 33270162
- [Background] Sassine J, Khawaja F, Shigle TL, Handy V, Foolad F, Aitken SL, Jiang Y, Champlin R, Shpall E, Rezvani K, Ariza-Heredia EJ, Chemaly RF. Refractory and Resistant Cytomegalovirus After Hematopoietic Cell Transplant in the Letermovir Primary Prophylaxis Era. Clin Infect Dis. 2021 Oct 20;73(8):1346-1354. doi: 10.1093/cid/ciab298. PMID 33830182